CLINICAL TRIAL: NCT00151697
Title: New Approach to Treat Type II Diabetes Failing on Maximal Oral Treatment
Brief Title: LANN-study: Lantus, Amaryl, Novorapid, Novomix Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTC 297-161104
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus Type II
Keywords: diabetes; failing oral treatment; weight gain
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Weight Gain | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart; glimepiride; Insulin Glargine

INTERVENTIONS:
Drug: Novomix 30
Drug: Novorapid and Amaryl
Drug: Lantus

SUMMARY:
Many diabetics gain weight while on insulin therapy. In this study, we evaluate the efficacy of the combination of glimepiride and short-acting insulin on weight control and glucose control. In this study, 150 diabetics whose diabetic control is inadequate while on maximal oral treatment will be randomized to either the new combination treatment or twice daily injections with a mixture of short- and longacting insulin or once-daily injection with a basal insulin analog. The study will compare glucose control and weight gain during a year after randomisation between the three treatments.

DETAILED DESCRIPTION:
Diabetic patients failing on maximal oral treatment usually switch to twice daily administration of a mixture of short- and longacting insulin. Although this improves glycemic control, it is generally accompanied by a substantial gain in body weight. This may lead to an increase in body fat resulting in a worsening of insulin resistance, leading to an increase in insulin dose needed to maintain glycemic control.

The combination of glimepiride(amaryl) and short-acting insulin (novorapid) is thought to attain glycemic control with a smaller increase in body weight.

In this randomized controlled trial, 150 diabetics failing on maximal oral treatment will be randomized to preprandial use of Novorapid combined with Amaryl at 20.00 hours, twice daily Novomix 30, or once daily Lantus. Metformin will be continued.

In the year after randomisation, patients will be followed for glycemic control, body weight, body composition, recorded number of hypoglycemic events, plasma lipid levels, basal and stimulated C-peptide levels and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* failing maximal oral treatment, defined as mean fasting blood glucose over 8 mmol/l and HbA1C over 7.5% for three months or more
* BMI 25 - 35 kg/m2
* fasting plasma C-peptide level over 0.3 nmol/l
* stable metformin and sulfonylurea dose for at least three months
* stable weight for at least three months (change maximal 2 kg)

Exclusion Criteria:

* fasting glucose over 25 mmol/l
* use of alpha-glucosidase inhibitors or thiazolidinediones in the two months preceding the study
* renal or liver failure defined as serum creatinine over 150 micromol/l, liver enzymes over 1.5 upper normal limit
* heart failure
* pregnancy
* alcohol more than two units per day
* inflammatory or infectious diseases
* unstable chronic disease
* discontinuation of smoking within three months of randomisation date
* allergy for or intolerance of glimepiride or novorapid.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-05

PRIMARY OUTCOMES:
glycemic control based on HbA1c
Body weight

SECONDARY OUTCOMES:
8-point glucose day curve of three consecutive days
24-hour glycemic control measured by continuous glucose monitoring for three consecutive days
recorded number of hypoglycemic events per month
waist circumference
dexa measurements of body composition
plasma lipid levels
basal and stimulated C-peptide levels
adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Hans de Boer, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

REFERENCES:
- [Background] de Boer H, Jansen M, Koerts J, Verschoor L. Prevention of weight gain in type 2 diabetes requiring insulin treatment. Diabetes Obes Metab. 2004 Mar;6(2):114-9. doi: 10.1111/j.1463-1326.2004.00322.x. PMID 14746576